CLINICAL TRIAL: NCT06372496
Title: A Phase 4, 52-week (Primary Analysis at 24-weeks), Randomized, Stratified, Open-label, Active-controlled, Parallel-group, Effectiveness Study, Comparing FF/UMEC/VI With Non-ellipta Usual Care (ICS/LABA) in Adult Participants With Uncontrolled Asthma
Brief Title: Pragmatic Open - Label Randomized Clinical Trial of FF/UMEC/VI vs Non-ellipta Usual Care ICS-LABA for Adult Participants With Uncontrolled Asthma
Acronym: PERFORM
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 219912
Record Dates: First submitted 2024-04-15; First posted 2024-04-18 (Actual); Last update posted 2025-10-22 (Actual); Status verified 2025-10

CONDITIONS: Asthma
Keywords: Asthma; FF/UMEC/VI; ICS/LABA
MeSH Terms: conditions — Asthma | interventions — fluticasone furoate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Fluticasone furoate/umeclidinium bromide/vilanterol trifenatate (FF/UMEC/VI) (Experimental)
  Interventions: Drug: Fluticasone furoate/umeclidinium bromide/vilanterol trifenatate
- Inhaled corticosteroids/long-acting beta-2 agonists (ICS/LABA) (Active Comparator)
  Interventions: Drug: Inhaled corticosteroids/long-acting beta-2 agonists

INTERVENTIONS:
Drug: Fluticasone furoate/umeclidinium bromide/vilanterol trifenatate — Participants will receive FF/UMEC/VI
  Arms: Fluticasone furoate/umeclidinium bromide/vilanterol trifenatate (FF/UMEC/VI)
Drug: Inhaled corticosteroids/long-acting beta-2 agonists — Participants will receive ICS/LABA
  Arms: Inhaled corticosteroids/long-acting beta-2 agonists (ICS/LABA)

SUMMARY:
The goal of this study is to assess and compare the effectiveness of fluticasone furoate/umeclidinium bromide/vilanterol trifenatate (FF/UMEC/VI) with inhaled corticosteroids/long-acting beta-2 agonists (ICS/LABA) in adult participants with uncontrolled asthma

ELIGIBILITY:
Inclusion Criteria:

Participants are eligible to be included in the study only if all of the following criteria apply:

1. Has a diagnosis of asthma as defined by Global Initiative for Asthma (GINA) 2023 guidelines for at least 3 months prior to randomization.
2. Participants who are either:

   * Currently untreated
   * Treated with daily maintenance ICS or ICS/LABA
3. ACQ-6 score ≥1.5 at randomization.
4. Participants able to perform technically acceptable and repeatable FEV1 maneuvers (i.e., a minimum of 2 acceptable and 1 repeatable effort) at visit 2 (V2)
5. Participants must be able to complete the study questionnaires.

Exclusion Criteria:

Participants are excluded from the study if any of the following criteria apply:

1. Recent history of life-threatening asthma
2. History of >1 severe exacerbation of asthma within 12 months prior to randomization.
3. Women of childbearing potential that are not following at least one highly effective method of contraception. This includes women who are pregnant or lactating or are planning on becoming pregnant during the study.
4. A WOCBP must have a negative pregnancy test ≤7 days prior to randomization.
5. Exposure to inhaler triple therapy [ICS + Long-acting muscarinic antagonist (LAMA) + LABA as Single inhaler triple therapy (SITT) or Multiple inhaler triple therapy(MITT)] and/or any LAMA-containing therapy within 12 months prior to randomization.
6. Ongoing need for biologic therapy or recent use of a biologic therapy
7. Participants with the diagnosis of chronic obstructive pulmonary disease, as per Global Initiative for Chronic Obstructive Lung Disease (GOLD 2024) guidelines.
8. Participants whose current medications include RELVAR ELLIPTA and ARNUITY ELLIPTA are not eligible to enter the study.
9. Participants who are medically unable to withhold their albuterol/salbutamol for 6 hours prior to spirometry testing
10. Changes in asthma medication (e.g., maintenance ICS/LABA) within 3 months prior to randomization.
11. Participants with a history of hypersensitivity to any of the study medications

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1357 (Actual)
Dates: Start 2024-04-16 (Actual); Primary Completion 2025-09-08 (Actual); Study Completion 2026-01-22 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in trough forced expiratory volume in 1 second (FEV1) | Baseline (Day 1), and at Week 24

SECONDARY OUTCOMES:
Number of participants achieving ≥0.5 point improvement from baseline for the Asthma Control Questionnaire-7 (ACQ-7) after 24 weeks of treatment | Baseline (Day 1), and Week 24
  The ACQ-7 consists of 7 questions scored between zero (no impairment/ limitation) to 6 (total impairment/ limitation).Higher scores indicate greater impairment. ACQ-7 is the responder analysis based on a 0.5 point change.
Number of participants achieving the composite endpoint (optimized) after 52 weeks of treatment | Up to 52 weeks
  The 4-point composite endpoint is defined as meeting the following criteria:
  * Change from baseline in trough FEV1 ≥ 100 mL at Week 52.
  * Controlled asthma based on ACQ-5 total score ≤ 1.5 at Week 52.
  * No severe asthma exacerbations over 52 weeks.
  * OCS-free over 52 weeks
Change from baseline in trough forced expiratory volume in 1 second (FEV1) after 52 weeks of treatment | Baseline (Day 1), and Week 52
Change from baseline in trough FEV1 ≥ 100mL after 24 and 52 weeks of treatment | Baseline (Day 1), Week 24 and Week 52
Change from baseline in through FEV1 ≥ 0mL after 24 and 52 weeks of treatment | Baseline (Day 1), Week 24 and Week 52
Number of participants achieving ≥0.5 point improvement from baseline for the ACQ-7 after 52 weeks of treatment | Week 52
  The ACQ-7 consists of 7 questions scored between zero (no impairment/ limitation) to 6 (total impairment/ limitation). Higher scores indicate greater impairment. ACQ-7 is the responder analysis based on a 0.5 point change.
Number of participants achieving ≥0.5 point improvement from baseline for the Asthma Control Questionnaire-6 (ACQ-6) after 24 and 52 weeks of treatment | Baseline (Day 1), Week 24 and Week 52
  The ACQ-6 is a shortened version of the ACQ-7 derived by removing one element (lung function element) from the original version. The scoring ranges from 0 (no impairment/ limitation) to 6 (total impairment/ limitation), higher scores indicate greater impairment. ACQ-6 is the responder analysis based on a 0.5 point change.
Number of participants achieving ≥0.5 point improvement from baseline for the ACQ-5 after 24 and 52 weeks of treatment | Baseline (Day 1), Week 24 and Week 52
  The ACQ-5 consists of 5 questions scored from zero (no impairment/limitation) to six (total impairment/ limitation). Higher scores indicate greater impairment. It is a shorter version of ACQ-7 derived by removal of two elements (lung function and rescue use elements) from original version (ACQ-7). ACQ-5 is the responder analysis based on a 0.5 point change.
Change from baseline in the ACQ-7 total score after 24 and 52 weeks of treatment | Baseline (Day 1), Week 24 and Week 52
  The ACQ-7 total consists of 7 questions scored between zero (no impairment/ limitation) to 6 (total impairment/ limitation). Higher scores indicate greater impairment.
Change from baseline in the ACQ-5 total score after 24 and 52 weeks of treatment | Baseline (Day 1), Week 24 and Week 52
  The ACQ-5 total consists of 5 questions scored from zero (no impairment/limitation) to six (total impairment/ limitation). Higher scores indicate greater impairment. It is a shorter version of ACQ-7 derived by removal of two elements (lung function and rescue use elements) from original version (ACQ-7).
Change from baseline in the ACQ-6 total score after 24 and 52 weeks of treatment | Baseline (Day 1), Week 24 and Week 52
  The ACQ-6 total is a shortened version of the ACQ-7 derived by removing one element (lung function element) from the original version. The scoring ranges from 0 (no impairment/limitation) to 6 (total impairment/ limitation), higher scores indicate greater impairment.
Change from baseline in the Asthma Control Test (ACT) score after 24 and 52 weeks of treatment | Baseline (Day 1), Week 24 and Week 52
  The ACT is a 5-question health survey used to measure asthma control in participants aged ≥12 years. Each question is scored from 1 to 5 for a total score ranging from 5 to 25; with higher scores indicating better asthma control.
Number of participants achieving the composite endpoint among those on ICS/LABA prior to randomization | Week 52
  The 4-point composite endpoint is defined as meeting the following criteria:
  * Change from baseline in trough FEV1 ≥ 100 mL at Week 52
  * Controlled asthma based on ACQ-5 total score ≤ 1.5 at Week 52
  * No severe asthma exacerbations over 52 weeks
  * OCS-free over 52 weeks
Number of participants achieving the composite endpoint among those on no treatment prior to randomization | Up to 52 weeks
  The 4-point composite endpoint is defined as meeting the following criteria:
  * Change from baseline in trough FEV1 ≥ 100 mL at Week 52.
  * Controlled asthma based on ACQ-5 total score ≤ 1.5 at Week 52.
  * No severe asthma exacerbations over 52 weeks.
  * OCS-free over 52 weeks
Change from baseline in the Asthma Quality of Life Questionnaire (AQLQ-12) total scores after 24 and 52 weeks of treatment | Baseline (Day 1), Week 24 and Week 52
  The AQLQ (+12), is a modified version of the original AQLQ with standardized activities. The response scale ranges from 1 (totally impaired) to 7 (not at all impaired). The total score is the score from all 32 questions.
Change from baseline in the Asthma Quality of Life Questionnaire (AQLQ-12) domain scores after 24 and 52 weeks of treatment | Baseline (Day 1), Week 24 and Week 52
  The AQLQ (+12), is a modified version of the original AQLQ with standardized activities. The response scale ranges from 1 (totally impaired) to 7 (not at all impaired). The domain score looks at each domain individually - symptoms, activity limitation, emotional function and environmental stimuli.
Change from baseline in the four domains of the asthma-specific adaptation of the Work Productivity and Activity Impairment Questionnaire (WPAI:Asthma) after 24 and 52 weeks of treatment | Baseline (Day 1), Week 24 and Week 52
  WPAI is a self-administered tool to determine the degree to which asthma affected work productivity while at work and affected activities outside of work in the last 7 days. The WPAI questionnaire score represents the percentage of impairment, from 0 to 100%. Higher WPAI scores indicate greater activity impairment.
Change from baseline in trough forced expiratory volume in 1 second (FEV1) among participants on budesonide/formoterol prior to randomization | Baseline (Day 1), and Week 24
Number of participants achieving ≥0.5 points improvement from baseline for ACQ-7 among participants on ICS/LABA prior to randomization | Baseline (Day 1), Week 24 and Week 52
  The ACQ-7 consists of 7 questions scored between zero (no impairment/ limitation) to 6 (total impairment/ limitation). Higher scores indicate greater impairment. ACQ-7 is the responder analysis based on a 0.5 point change.
Change from baseline in the ACQ-7 total score among participants on ICS/LABA prior to randomization | Baseline (Day 1), Week 24 and Week 52
  The ACQ-7 total consists of 7 questions scored between zero (no impairment/ limitation) to 6 (total impairment/ limitation). Higher scores indicate greater impairment.
Change from baseline in trough forced expiratory volume in 1 second (FEV1) for participants with no treatment prior to randomization. | Baseline (Day 1), and Week 24
Number of participants achieving ≥0.5 points improvement from baseline for ACQ-7 for participants with no treatment prior to randomization. | Baseline (Day 1), Week 24 and Week 52
  The ACQ-7 consists of 7 questions scored between zero (no impairment/ limitation) to 6 (total impairment/ limitation). Higher scores indicate greater impairment. ACQ-7 is the responder analysis based on a 0.5 point change.
Change from baseline in the ACQ-7 total score for participants with no treatment prior to randomization. | Baseline (Day 1), Week 24 and Week 52
  The ACQ-7 total consists of 7 questions scored between zero (no impairment/ limitation) to 6 (total impairment/ limitation). Higher scores indicate greater impairment. s

CONTACTS AND LOCATIONS:
Locations (59):
- United States (25):
  - GSK Investigational Site, Little Rock, Arkansas
  - GSK Investigational Site, Newport Beach, California
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, North Miami Beach, Florida
  - GSK Investigational Site, Orlando, Florida
  - GSK Investigational Site, Palm Springs, Florida
  - GSK Investigational Site, Port Charlotte, Florida
  - GSK Investigational Site, Tallahassee, Florida
  - GSK Investigational Site, Normal, Illinois
  - GSK Investigational Site, New Orleans, Louisiana
  - GSK Investigational Site, Bangor, Maine
  - GSK Investigational Site, Warren, Michigan
  - GSK Investigational Site, Missoula, Montana
  - GSK Investigational Site, Papillion, Nebraska
  - GSK Investigational Site, Linwood, New Jersey
  - GSK Investigational Site, New Windsor, New York
  - GSK Investigational Site, Asheville, North Carolina
  - GSK Investigational Site, Charlotte, North Carolina
  - GSK Investigational Site, Cincinnati, Ohio
  - GSK Investigational Site, Philadelphia, Pennsylvania
  - GSK Investigational Site, Pittsburgh, Pennsylvania
  - GSK Investigational Site, Rock Hill, South Carolina
  - GSK Investigational Site, Spartanburg, South Carolina
  - GSK Investigational Site, Beaumont, Texas
  - GSK Investigational Site, Dallas, Texas
- Argentina (5):
  - GSK Investigational Site, Buenos Aires
  - GSK Investigational Site, Concepción del Uruguay
  - GSK Investigational Site, Mendoza
  - GSK Investigational Site, Quilmes
  - GSK Investigational Site, Rosario
- Australia (8):
  - GSK Investigational Site, Bruce, Australian Capital Territory
  - GSK Investigational Site, Blacktown, New South Wales
  - GSK Investigational Site, Coffs Harbour, New South Wales
  - GSK Investigational Site, Kanwal, New South Wales
  - GSK Investigational Site, Sydney, New South Wales
  - GSK Investigational Site, Brisbane, Queensland
  - GSK Investigational Site, Osborne Park, Western Australia
  - GSK Investigational Site, Spearwood, Western Australia
- Canada (2):
  - GSK Investigational Site, Windsor, Ontario
  - GSK Investigational Site, Trois-Rivières, Quebec
- Japan (16):
  - GSK Investigational Site, Fukuoka
  - GSK Investigational Site, Gifu
  - GSK Investigational Site, Hiroshima
  - GSK Investigational Site, Hyōgo
  - GSK Investigational Site, Kagawa
  - GSK Investigational Site, Kagoshima
  - GSK Investigational Site, Kanagawa
  - GSK Investigational Site, Kumamoto
  - GSK Investigational Site, Matsuyama
  - GSK Investigational Site, Miyazaki
  - GSK Investigational Site, Nagaoka-Shi
  - GSK Investigational Site, Niigata
  - GSK Investigational Site, Okawa-shi
  - GSK Investigational Site, Ōita
  - GSK Investigational Site, Tokyo
  - GSK Investigational Site, Yokohama
- GSK Investigational Site, Seoul, South Korea
- Taiwan (2):
  - GSK Investigational Site, Kaohsiung City
  - GSK Investigational Site, Taichung

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to anonymized individual patient-level data (IPD) and related study documents of the eligible studies via the Data Sharing Portal. Details on GSK's data sharing criteria can be found at: https://www.gsk.com/en-gb/innovation/trials/data-transparency/
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Anonymized IPD will be made available within 6 months of publication of primary, key secondary and safety results for studies in product with approved indication(s) or terminated asset(s) across all indications.
Access Criteria: Anonymized IPD is shared with researchers whose proposals are approved by an Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension may be granted, when justified, for up to 6 months.
URL: https://www.gsk.com/en-gb/innovation/trials/data-transparency/